CLINICAL TRIAL: NCT06568770
Title: Comparison of Ease of SPINAL Positioning Between USG Guided Supra-inguinal Fascia Iliaca Block vs USG Guided Pericapsular Nerve Group Block in Patients Undergoing Femur Fracture Surgery
Brief Title: Comparison of EOSP Between Usg Guided S-FICB vs USG Guided PENG Block in Pts Undergoing Femur Fracture Surgery
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sahiwal medical college sahiwal (Other Government)
Responsible Party: Principal Investigator, Shajeea Asghar, Resident Anaesthetist, District Headquarters Teaching Hospital Sahiwal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 211/IRB
Record Dates: First submitted 2024-08-13; First posted 2024-08-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Post Operative Pain; Bradycardia; Hypotension; Femur Fracture
Keywords: PENG,S-FICB,ASA,EOSP
MeSH Terms: conditions — Pain, Postoperative; Bradycardia; Hypotension; Femoral Fractures

STUDY DESIGN:
Intervention Model Description: Group 1 will receive S-FICB and Group 2 will receive PENG
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GROUP S-FICB (Other): Suprainguinal Facia iliaca Block
  Interventions: Drug: USG GUIDED SUPRA-INGUINAL FASCIA ILIACA BLOCK
- GROUP-PENG (Other): Pericapsular Nerve Group Block
  Interventions: Drug: PERICAPSULAR NERVE BLOCK

INTERVENTIONS:
Drug: USG GUIDED SUPRA-INGUINAL FASCIA ILIACA BLOCK — With the patient in the proper position, the skin will be disinfected and the transducer positioned to identify the femoral artery and the iliopsoas muscle and fascia iliaca. The transducer will be moved laterally until the sartorius muscle is identified. As the needle will eventually pierce the fascia, maybe a "pop" will be felt. After negative aspiration, 1-2 mL of local anesthetic will be injected to confirm the proper injection plane between the fascia and the ilio-psoas muscle. A proper injection will result in the separation of the fascia iliaca by the local anesthetic in the medial-lateral direction from the point of injection as described. After the spread of the drug will be seen, the rest of the drug volume will be injected
  Other Names: S-FICB
  Arms: GROUP S-FICB
Drug: PERICAPSULAR NERVE BLOCK — an ultrasound probe will be placed over the line joining anterior superior iliac spine (ASIS) and pubic tubercle (PT) keeping lateral margin at ASIS and adjusted the probe to get a sonoanatomic view for PENG block. The needle entry point will be selected on the skin in such a manner that perpendicular needle entry will guide needle near target point iliopectineal eminence (IPE). The needle entry point will be anaesthetized with 2 ml 1% lidocaine and 22G 80mm stimuplex needle will be inserted "out-of- plane" to reach the bony rim near IPE avoiding injury to femoral nerve (visible just lateral to femoral artery). On bony contact, 20 ml 0.5% bupivacaine will be injected slowly with repeated aspiration to avoid intravascular injection. The correct needle position will be confirmed by drug spread under ilio-psoas muscle and then the rest of the drug volume will be injected.
  Other Names: PENG
  Arms: GROUP-PENG

SUMMARY:
To compare the immediate and postoperative analgesic efficacy of S-FICB and PENG block will be the objective. The use of ultrasonography in anesthesia has helped the anesthetist to see the nerve, needle and the distribution of the drug, thereby enhancing the chances of a favorable outcome of the nerve block. Grade A recommendation for an ultrasound guided approach to the peripheral nerve blocks is supported by level Ib evidence for a shortened time for the onset of sensory block, decreased performance time and lower drug doses10.

Although individually both the blocks have been studied, there are only a handful of studies comparing both techniques under ultrasound guidance for making patient positioning for spinal anesthesia easy. And no local data is available comparing these blocks. So, we want to compare the analgesic efficacy of USG PENG block with USG S-FICB block in patients with fracture femur in reducing pain associated with positioning (sitting) for subarachnoid block, duration of analgesia, opioid sparing effect and complications. So that procedure with better analgesic efficacy and less complications will be included in our local guidelines as a part of multimodal analgesia.

DETAILED DESCRIPTION:
Patients fulfilling the inclusion criteria will be included. Patients will be optimized for dressing. A detailed history will be taken regarding the mode of injury, any pre-existing disease and previous surgery followed by the local examination of the patient will be done to rule out any systemic disease. Informed consent will be taken. These patients will be divided into 2 groups by Computer-generated random numbers and group assignment will be done by sequentially numbered opaque envelopes. The envelope will be opened just before the procedure by the anaesthesiologist performing the block. The observer (another anaesthesiologist) and patients will be unaware of the group and procedure performed. Group A (Supra-inguinal Fascia Iliaca Block) and Group B (Pericapsular Nerve Group Block). The monitors of electrocardiogram, pulse oximetry and non-invasive blood pressure in the preoperative area will be connected. For drug and fluid administration, an intravenous cannula of suitable size will be obtained. Pre-procedural pain will be assessed during rest as well as on movement (15° passive elevation) of the affected limb and will be recorded on numeric pain rating scale (NRS) [0 = no pain; 10 = worst imaginable pain]. The blocks will be performed in supine position and strict sterile technique will be followed. Both the blocks will be performed as per the standard technique. The site to be blocked will be painted with 5% povidone-iodine followed by spirit and will be draped. A linear 7-13 MHz ultrasonography probe (ACUSON P500, digital colour doppler ultrasound, Siemens Germany) will be used with in-plane approach of needle. Group S-FIB (n = 35, those who will receive a S-FIB with 20 mL of 0.5% bupivacaine) and group PENG (n = 35, those who will receive a PENG with 20 mL of 0.5% bupivacaine). Depending on the allotted group, patients will be given the block under the guidance of ultrasound in the preoperative area by an experienced anesthesiologist with more than two years' experience. The PENG block will be performed as follows: an ultrasound probe will be placed over the line joining anterior superior iliac spine (ASIS) and pubic tubercle (PT) keeping lateral margin at ASIS and adjusted the probe to get a sonoanatomic view for PENG block. The needle entry point will be selected on the skin in such a manner that perpendicular needle entry will guide needle near target point iliopectineal eminence (IPE). The needle entry point will be anaesthetized with 2 ml 1% lidocaine and 22G 80mm stimuplex needle will be inserted "out-of- plane" to reach the bony rim near IPE avoiding injury to femoral nerve (visible just lateral to femoral artery). On bony contact, 20 ml 0.5% bupivacaine will be injected slowly with repeated aspiration to avoid intravascular injection. The correct needle position will be confirmed by drug spread under ilio-psoas muscle and then the rest of the drug volume will be injected. The S-FIB will be given in a similar fashion. With the patient in the proper position, the skin will be disinfected and the transducer positioned to identify the femoral artery and the iliopsoas muscle and fascia iliaca. The transducer will be moved laterally until the sartorius muscle is identified. As the needle will eventually pierce the fascia, maybe a "pop" will be felt. After negative aspiration, 1-2 mL of local anesthetic will be injected to confirm the proper injection plane between the fascia and the ilio-psoas muscle. A proper injection will result in the separation of the fascia iliaca by the local anesthetic in the medial-lateral direction from the point of injection as described. After the spread of the drug will be seen, the rest of the drug volume will be injected. A numerical rating scale (NRS) pain score will be recorded before the block. The onset time to achieve NRS pain score of 4 or less than 4 will be noted on prescribed proforma for both groups. The patients will be made to sit for spinal anesthesia when the NRS score will be less than 4 after preloading with ringer lactate solution @80ml/kg. The spinal anaesthesia will be performed using 25G spinal needle () with 0.75% bupivacaine solution (2ml) in both groups. The monitors of electrocardiogram, pulse oximetry, non-invasive blood pressure and urine output will be monitored according to ASA standard. After completion of surgery patient will be shifted to respective ward where trained doctor and staff will monitor the patient. The NRS score will be measured immediately postoperatively and at intervals of 2 hours for a period of 24 hours. If the NRS score will be > 4, rescue analgesia will be given; an injection of paracetamol 15 mg/kg will be given over a period of 10 to 15 minutes as an intravenous infusion and time will be noted. Inj nalbuphine 0.1mg/kg will be given for breakthrough pain. Total dose of intravenous nalbuphine will be recorded in 1st 24hrs.

ELIGIBILITY:
Inclusion Criteria:

* 1. Both Genders (Male /Female). 2. Age between 20 years to 70 years. 3. Radiologically confirmed femur fracture. 4. ASA Class I, II, III.

Exclusion Criteria:

1. Patient refusal
2. Other distracting painful pathology
3. Any contraindication to Spinal Anesthesia or peripheral nerve blocks
4. Coagulopathic disorders
5. H/O ischemic heart disease
6. Patients on opioids for chronic pain
7. Patients with significant cognitive impairment
8. Patients with no pain while sitting by themselves without any support.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Ease Of Spinal Positioning | 20 minutes till Performance of spinal anaesthesia
  The ease of spinal positioning (EOSP) will be assessed on the scale of 0-3 0 = unable to position
  1. = patient had abnormal posturing due to pain and required support for positioning
  2. = mild discomfort but does not require support for positioning
  3. = optimal condition where the patient was able to position himself without pain

SECONDARY OUTCOMES:
Post op Analgesia | from performance of block to first rescue analgesia(in hours)
  Duration of post op analgesia.
opioid sparing effect | 24 hrs
  total opioid consumption in mg/24hrs

OTHER OUTCOMES:
Post op Nausea Vomiting | 24 hrs
  Post Op Nausea Vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Riaz, MD, Study Director — Sahiwal medical college sahiwal
Locations (1):
- Sahiwal Medical College, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request after completion of study i.e. March 2025.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: March 2025
Access Criteria: On Demand